CLINICAL TRIAL: NCT02999438
Title: Frailty in Children With Cardiac Disease: A Pilot Study
Brief Title: Frailty in Children With Cardiac Disease
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Brian Birnbaum, Physician, Associate Professor of Pediatrics, Children's Mercy Hospital Kansas City
Other Study IDs: 16060468
Record Dates: First submitted 2016-12-19; First posted 2016-12-21 (Estimated); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Pulmonary Hypertension; Heart Failure; Single Ventricle
MeSH Terms: conditions — Hypertension, Pulmonary; Heart Failure; Univentricular Heart

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with hemodynamically significant heart disease: Patients with either:
  1. Single ventricle physiology s/p Fontan
  2. Heart failure diagnosed by a cardiologist
  3. Pulmonary hypertension diagnosed by cath
  Interventions: Device: Actigraph to check activity levels at home
- Controls: Healthy controls as defined in inclusion- exclusion criteria
  Interventions: Device: Actigraph to check activity levels at home

INTERVENTIONS:
Device: Actigraph to check activity levels at home

SUMMARY:
Frailty is a complex biologic syndrome of diminished physiologic reserve that leads to decreased resistance to stressors and is associated with adverse health outcomes. The syndrome has been well studied in adults and is quantified by the Fried criteria, which are comprised of five components- slowness, weakness, self-reported exhaustion, shrinkage and diminished physical activity. The concept of frailty is novel in children. A study in young adult childhood cancer survivors demonstrated increased incidence of frailty in this population along with increased risk of morbidity and mortality. This suggests that frailty as a phenotype has relevance outside of the geriatric age group. Pediatric patients with single ventricle physiology, heart failure and pulmonary artery hypertension- all represent populations with significantly increased risk of mortality, morbidity and decreased quality of life. Currently, such patients are monitored outpatient by serial echocardiograms and blood work that only gives information about end organ damage. But there is no validated tool available to measure global infirmity in such children. Better understanding of the relevance and applicability of frailty in pediatrics may allow for identification of the most vulnerable pediatric cardiac patients and be of value in optimizing their clinical management and improving health outcomes.

ELIGIBILITY:
Inclusion Criteria:

SUBJECT/CASE POPULATION herein referred to as Subjects:

* Children and adolescents between the ages of 8.0-17.50 years
* Subjects must be diagnosed with one of the following heart conditions:

  * Subjects with single ventricle physiology and Fontan surgery completion at least 6 months prior to study enrollment
  * Subjects with diagnosis of heart failure by a cardiologist
  * Subjects with a diagnosis of pulmonary arterial hypertension, confirmed by cardiac catheterization, requiring use of at least 1 pulmonary vasodilator or oxygen for their pulmonary hypertension

CONTROL POPULATION herein referred to as Controls:

* Healthy children and adolescents between the ages of 8.0-17.50 years

Exclusion Criteria:

BOTH SUBJECT/CASE POPULATION AND CONTROL POPULATION:

* Subjects or controls with known severe neurological or respiratory diseases, eating disorders (such as anorexia, bulimia) or physical limitations (wheelchair bound) which may impact their ability to perform study procedures in the opinion of the provider.
* Subjects or controls with tracheostomy and ventilator dependency
* Subjects or controls with unstable angina/ myocardial infarction in the last 4 weeks
* Subjects or controls who are unable to perform 6 continuous minutes of walking, hand-grip dynamometry, or complete questionnaire measures as described.

SUBJECT/ CASE POPULATION:

* Subjects with heart transplantation within the past 1 year
* Subject will be excluded if the cardiologist feels that the study is not appropriate for the subject.

CONTROL POPULATION:

* Controls with any known chronic medical condition requiring some medication over the past 30 days.
* Controls on any chronic prescription medicines for > 30 days

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The investigators are studying children with single ventricle physiology, s/p Fontan, patients with heart failure and pulmonary hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2016-11; Primary Completion 2022-09 (Actual); Study Completion 2022-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Frailty in children with hemodynamically significant heart disease | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Brian Birnbaum, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

REFERENCES:
- [Derived] Panchangam C, White DA, Goudar S, Birnbaum B, Malloy-Walton L, Gross-Toalson J, Reid KJ, Shirali G, Parthiban A. Translation of the Frailty Paradigm from Older Adults to Children with Cardiac Disease. Pediatr Cardiol. 2020 Jun;41(5):1031-1041. doi: 10.1007/s00246-020-02354-7. Epub 2020 May 6. PMID 32377892